CLINICAL TRIAL: NCT04431804
Title: Effect of Thyme and Carvacroll Nanoparticles on Aspergillus Fumigatus Isolate From Intensive Care Patients
Brief Title: THYME AND CARVACROLL Nanoparticle Effect on Fungi
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anaesthesia, Assiut University
Other Study IDs: wwww
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Aspergillosis
MeSH Terms: conditions — Aspergillosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: silver nanoparticle — fungicidal effect of silver nanoparticles on aspergillus isolates

SUMMARY:
Invasive Aspergillosis (IA) has increasingly been recognized as an emerging disease of non-neutropenic patients and in patients admitted to the ICU, even in the absence of an apparent predisposing immune-deficiency, with incidence ranges from 0.3% to 5.8% with an overall mortality rate exceeding 80%.

ELIGIBILITY:
Inclusion Criteria:

* intensive care patients

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: intensive care patients
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
fungicidal effect of silver nanoparticles on aspergillus fumigatus | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt